CLINICAL TRIAL: NCT02857088
Title: Study of the Emotional Reactivity to Olfactive and Visual Perception in Depressed Patients
Brief Title: Olfactory and Visual Perception in Depressed Patients
Acronym: PERODEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unavailable recording device and difficulty of patient inclusions
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P/2011/126
Record Dates: First submitted 2016-07-26; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Depression
Keywords: depression; emotional reactivity
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- depressed patients (Experimental): patient with a current unipolar major depressive disorder intervention: olfactory assessment, image visualization and psychophysiological assessment
  Interventions: Behavioral: olfactory assessment; Behavioral: image visualization; Behavioral: psychophysiological assessment
- non depressed subject (Experimental): subject without a current unipolar major depressive disorder intervention: olfactory assessment, image visualization and psychophysiological assessment
  Interventions: Behavioral: olfactory assessment; Behavioral: image visualization; Behavioral: psychophysiological assessment

INTERVENTIONS:
Behavioral: olfactory assessment — determination of olfactory sensitivity through olfactory threshold assessment (butanol) determination of hedonicity and intensity of 16 usual odors
Behavioral: image visualization — 20 images (from the IAPS-international affective picture systems) are presented to the subject. He has to determine the hedonicity of each picture.
Behavioral: psychophysiological assessment — during the olfaction assessment and the image visualization, skin conductance reactivity (SCR) is recorded to assess unconscious emotional reactivity

SUMMARY:
The study aimed to determine the emotional reactivity of depressed patients to visual and olfactory stimuli in comparison with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* no cognitive impairment that could prevent instruction comprehension
* no more than 10 cigarettes/day
* signed informed consent
* group 1: current major depressive disorder
* group 2: no current major depressive disorder

Exclusion Criteria:

* pregnancy
* visual impairment
* olfactory impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
hedonicity score of visual stimuli | up to 1 month
  it will be compared between depressed and non depressed subjects.
skin conductance reactivity amplitude | up to 1 month
  it will be compared between depressed and non depressed subjects.
Skin conductance reactivity reaction time | up to 1 month
  it will be compared between depressed and non depressed subjects.
hedonicity score of olfactory stimuli | up to 1 month
  it will be compared between depressed and non depressed subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Nezelof, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No